CLINICAL TRIAL: NCT02249689
Title: Three-month Clinical Evaluation of Silicone Hydrogel Definitive 65 Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contamac Ltd (Industry)
Collaborators: Hartwig Research Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-001-001
Record Dates: First submitted 2014-01-19; First posted 2014-09-25 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive 65 (Experimental): The Test product were the Definitive 65 (Filcon V4) lenses. This material is produced by Contamac Ltd. and the contact lenses were manufactured by Appenzeller Kontaktlinsen AG.
  Interventions: Other: Definitive 65
- Definitive 74 (Active Comparator): The Control product was the commercially available Definitive 74 (Efrofilcon A) lens. This material is produced by Contamac Ltd. and the contact lenses were manufactured by Appenzeller Kontaktlinsen AG.
  Interventions: Other: Definitive 74

INTERVENTIONS:
Other: Definitive 65
  Arms: Definitive 65
Other: Definitive 74
  Arms: Definitive 74

SUMMARY:
Comparison of different contact lens materials.

DETAILED DESCRIPTION:
This will be a 3-month, open-label, bilateral, parallel-group, randomised, daily wear study. Two-thirds of the subjects will wear the Test lenses in both eyes, and one-third will wear the Control lenses in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to sign the informed consent form
* ages 18 years or older
* Subjects must have owned spectacles or contact lenses prior to enrolment for this trial
* spherical power between -10.00 D and +10.00 D (at vertex distance 0 mm)
* astigmatic power equal to or less than 0.75 D

Exclusion Criteria:

* eye injury or surgery within 3 months immediately prior to enrolment for this trial
* pre-existing ocular irritation that would preclude contact lens fitting
* currently enrolled in an ophthalmic clinical trial
* evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses use of as determined by the investigator
* any use of medications for which contact lens wear could be contradicted, as determined by the investigator
* current extended-wear users (sleep-in overnight)
* current monovision leans wearers
* pregnant women and nursing mothers
* best-corrected visual acuity worse than 6/9 (logMAR: +0.20; Snellen decimal: 0.63)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
questionnaire addressing subjective comfort and wear time | subjects will be followed-up for three months
  Subjects rated on a scale from 1 to 10, where 1 was 'poor' and 10 was 'excellent'.
limbal redness - ocular biomicroscopy | subjects will be followed-up for three months
  Findings were graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.
corneal staining - ocular biomicroscopy | subjects will be followed-up for three months
  Findings were graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartwig, PhD, Principal Investigator — Hartwig Research Center
Locations (2):
- Germany (2):
  - Siehste, Kassel
  - Kresinsky, Würzburg